CLINICAL TRIAL: NCT03098524
Title: Low Tidal MEChanical Ventilation Against NO Ventilation During Cardiopulmonary Bypass Heart Surgery : a Randomized Controlled Trial
Brief Title: Low Tidal MEChanical Ventilation Against NO Ventilation During Cardiopulmonary Bypass Heart Surgery
Acronym: MECANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016/03
Record Dates: First submitted 2017-02-27; First posted 2017-03-31 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Failure; Atelectasis; Pneumonia; Pneumothorax; Bleeding; Surgery--Complications; Cardiac Disease
Keywords: Cardiac surgery; Mechanical ventilation; Cardiopulmonary bypass; Pneumonia; Atelectasis
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Atelectasis; Pneumonia; Pneumothorax; Hemorrhage; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients are ventilated or not during the time they are sedated, so they are blind to their study arm.
  Anesthesiologists perform mechanical ventilation or not during cardiopulmonary bypass and log per-operative data (such as number of insufflations) on a separate leaflet of the eCRF. Investigators (cardiologists and critical care specialists) are not aware of the treatment arm as it is performed during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low tidal volume ventilation (LTV arm) (Experimental): During cardiopulmonary bypass, mechanical ventilation is maintained with 5 acts/minute, tidal volume = 3 ml/kg (ideal body weight) with positive end-expiratory pressure = 5 cmH2O
  Interventions: Procedure: Low tidal volume ventilation (LTV arm); Procedure: Lung recruitment manoeuver
- No ventilation (noV arm) (Placebo Comparator): No mechanical ventilation during cardiopulmonary bypass.
  Interventions: Procedure: No ventilation (noV arm); Procedure: Lung recruitment manoeuver

INTERVENTIONS:
Procedure: Low tidal volume ventilation (LTV arm) — During cardiopulmonary bypass, mechanical ventilation is maintained with settings described above.
  Arms: Low tidal volume ventilation (LTV arm)
Procedure: No ventilation (noV arm) — During cardiopulmonary bypass, no mechanical ventilation is performed.
  Arms: No ventilation (noV arm)
Procedure: Lung recruitment manoeuver — An insufflation with positive end-expiratory pressure +30 cmH20 during 5 seconds.
  At the end of cardiopulmonary bypass, in the operative room. And after transfer to the ICU (intensive care unit).

SUMMARY:
BACKGROUND. Postoperative pulmonary complications are a leading cause of morbidity and mortality after cardiac surgery. To this date, there are no recommendations regarding mechanical ventilation associated with cardiopulmonary bypass (CPB) during the surgery and anesthesiologists perform either no ventilation (noV) at all during CPB or maintain a low-tidal volume ventilation (LTV). Indirect evidence points towards better pulmonary outcomes when LTV is performed but no proper prospective trial with large inclusion of all types of cardiac surgery has been published.

DESIGN. The MECANO trial is a single-center, double-blind, randomized controlled trial comparing two mechanical ventilation strategies, noV and LTV, during cardiac surgery with CPB. 1500 patients will be included for whom planned cardiac surgery with CPB is performed. They will be randomized between noV and LTV, on a 1:1 ratio. The noV group will receive no ventilation during CPB. The LTV group will receive 5 acts/minute with a tidal volume of 3 mL/kg and positive end-expiratory pressure of 5 cmH2O. Primary endpoint will be composite of overall death, early respiratory failure defined as PaO2/FiO2 ratio <200 mmHg at one-hour after arrival in the ICU, heavy oxygenation support (defined as a patient requiring either non-invasive ventilation, mechanical ventilation or high flow oxygen) at 2 days after arrival in the ICU or ventilator acquired pneumoniae defined by Center of Disease Control. Lung recruitment manoeuvers will be performed for noV and LTV groups, at the end of surgery and at the arrival in ICU with an insufflation at +30 cmH20 during 5 seconds. Secondary endpoints are those composing the primary endpoint with the addition of pneumothorax, CPB duration, quantity of postoperative bleeding, red blood cells transfusions, revision surgery requirements, length of stay in the ICU and in the hospital and total hospitalization costs. Patients will be followed until hospital discharge.

SUMMARY. The MECANO trial compares a no-ventilation to a low-tidal volume strategy for mechanical ventilation during cardiac surgery with CPB, regarding a primary composite outcome including death, respiratory failure and pneumoniae.

DETAILED DESCRIPTION:
BACKGROUND. Ventilator-acquired pneumonia (VAP) are a common postoperative complication and account for a large part of post-cardiac surgery morbidity and mortality. Incidence of VAP depends on numerous factors, some of which are pulmonary collapsus and atelectasis during cardiopulmonary bypass, a lowering of bronchial arterial blood flow and a systemic inflammation response syndrome during and after cardiopulmonary bypass (CPB).

On the one hand, CPB allows blood oxygenation during cardiac surgery, regardless of heartbeat and oscillations, allowing surgeon to operate without disturbance.

On the other hand, postoperative pulmonary complications appear to be more frequent when no mechanical ventilation is maintained while under CPB.

Recent meta-analysis found oxygenation improvement after the weaning from CPB when low-tidal-volume (LTV) ventilation was maintained or after lung recruitment maneuvers (LRM), as compared to when there was no ventilation (noV). Furthermore, maintaining mechanical ventilation would reduce the inflammation response and tissue damage. The design of these studies did not provide with clinical hard endpoints such as respiratory complications, death or length of stay, hence, an unquestionable standardized strategy of lung protection during CPB has not been evidenced at this time and there are no scientific recommendations on whether mechanical ventilation has to be maintained during cardiac surgery or not, notably between low-tidal volume ventilation (LTV) and no-ventilation (noV).

The investigators aim to prove superiority of LTV over noV strategy during CPB in cardiac surgery, in order to decrease postoperative respiratory complications.

DESIGN. The MECANO trial is a single-center, double-blind, non-pharmacological, randomized controlled trial comparing two mechanical ventilation strategies, LTV and noV, during cardiac surgery with CPB.

Population. All patients aged more than 18 years will be eligible planned for cardiac surgery with CPB will be eligible. All patients will provide written informed consent before their inclusion in the trial.

Endpoints. Primary endpoint will be composite of overall death, early respiratory failure defined as PaO2/FiO2 ratio <200 at one-hour after arrival in the ICU, heavy oxygenation support (defined as a patient requiring either non-invasive ventilation, mechanical ventilation or high flow oxygen) at 2 days after arrival in the ICU or ventilator acquired pneumoniae defined by Center of Disease Control. Secondary endpoints are those composing the primary endpoint with the addition of pneumothorax, CPB duration, volume of postoperative bleeding, red blood cells transfusions, requirements for revision surgery, length of stay in the ICU and in the hospital and total hospitalization costs. Patients will be followed until hospital discharge.

Randomization. Patients will be randomized by the anesthesiologist when arriving in the operating room, between LTV and noV arm, on a 1:1 ratio, using a web software. Only the anesthesiologist will be aware of the allocation arm in order for him to perform the necessary ventilation strategy, however, physicians outside the operating room (hence, study investigators) will not be aware of the treatment arm. Any deviation from the protocol will be recorded, as will be the reason of deviation.

Intervention. The noV group will receive no ventilation during CPB. The LTV group will receive 5 acts/minute with a tidal volume of 3 mL/kg and positive end-expiratory pressure of 5 cmH2O.

Lung recruitment maneuvers will be performed in both groups, at the end of surgery, and at the arrival in ICU with insufflation at +30 cmH20 during 5 seconds. In ICU, ventilation strategy will be lung-protective with: tidal volume=6 ml/kg of ideal body weight, PEEP=5 cmH2O, FiO2 set to obtain PaO2 between 200 and 250 mmHg, inspiration/expiration time ratio = 1:2. Other therapeutics will be left to the appreciation of the critical care medicine specialist.

Data collection. All data will be recorded on a dedicated CRF. Preoperative data will be collected prior to the surgery (age, height, weight, Euroscore 2, smoking status, diabetes, peripheral arterial disease, pulmonary comorbidity, forced expiratory volume in one second, pulmonary infection in the past 30 days, creatininemia). Variables linked to the surgery will be: type of surgery, duration of CPB, number of red blood cells transfusions, number and reasons of manual insufflations. Daily visit will record temperature, PaO2, FiO2, ventilation mode, hemoglobinemia, leucocytemia, quantity of bleeding and any of the endpoints listed above. Time to events will be recorded as well. Follow up will be maintained until hospital discharge.

Statistical considerations Sample-size calculation was based on a two-sided alpha error of 0.05 and a 80% power. On the basis of respiratory insufficiency incidence after cardiac surgery, the investigators anticipate at least 25% of patients presenting postoperative respiratory complications. A relative improvement in the incidence of primary outcome of 20% between the 2 arms (odd-ratio 0.8 in favor of LTV arm as compared to noV arm) is expected. The required sample size is then 720 patients per group, 1440 patients in total. Accounting for attrition ratio, 1500 patients will be included. Intermediary analysis will be performed.

Data analysis. Patients will be analyzed following intention to treat principle. Logistic regression will be performed for statistical analysis. Relative risks with 95% confidence intervals and differences between medians with 95% confidence intervals will be calculated when appropriate. Two-sided significance tests will be used throughout. The investigators will infer a subgroup effect if the interaction term of treatment and subgroup is statistically significant at P <0.05.

ELIGIBILITY:
Inclusion:

more than 18 years old

ability to provide an informed consent

planned surgery

surgical intervention with cardio-pulmonary bypass, aortic clamp and cardioplegia.

Exclusion:

impossibility to wean CPB at the end of cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or early respiratory failure or Late respiratory failure or Ventilator acquired pneumonia and early pneumonia | From date of randomization until the date of first documented event or date of death from any cause, whichever came first, assessed up to 24 months.
  Composite outcome with all-cause in-hospital mortality, early respiratory failure defined as PaO2/FiO2 ratio <200 at the first hour after transfer in ICU after surgery, late respiratory failure defined as heavy oxygenation support (non-invasive ventilation, high flow oxygen or mechanical ventilation) two days after surgery and pneumonia (early or ventilator acquired) defined by Center of Disease Control (CDC) criteria (2016 guidelines).

SECONDARY OUTCOMES:
All-cause in-hospital mortality | From date of randomization until date of death from any cause, assessed up to 24 months.
  All-cause in-hospital mortality
Early respiratory failure | Assessed at one hour after transfer in postoperative ICU
  PaO2/FiO2 ratio <200 at the first hour after transfer in ICU after surgery
heavy oxygenation support | Assessed 2 days after surgery
  requirement of non-invasive ventilation, high flow oxygen or mechanical ventilation
Pneumonia (early or ventilator-acquired) | From date of randomization until the date of first documented event, assessed up to 24 months.
  pneumonia (early or ventilator acquired) defined by Center of Disease Control (CDC) criteria (2016 guidelines), diagnosed while in-hospital after the cardiac surgery.
Length of stay in the ICU | Assessed at the end of hospitalization, through study completion, assessed up to 24 months.
  Length of stay in the intensive care unit (ICU) (days) after the initial cardiac surgery
Length of stay in the hospital | Assessed at the end of hospitalization, through study completion, assessed up to 24 months.
  Length of stay in the hospital (days) after the initial cardiac surgery
Cost of hospitalization | Assessed at the end of hospitalization, through study completion, assessed up to 24 months.
  Cost of hospitalization (euros)

OTHER OUTCOMES:
Revision surgery | From date of randomization until the date of first documented event, assessed up to 24 months.
  Requirement for any revision cardiac surgery after the initial surgery
Pneumothorax | From date of randomization until the date of first documented event, assessed up to 24 months.
  Pneumothorax diagnosed on chest x-ray or TDM occurring after the initial surgery
Postoperative bleeding | Assessed at the end of hospitalization, through study completion, assessed up to 24 months.
  Postoperative bleeding (mL)
Cardiopulmonary bypass duration | Assessed at the end of the initial cardiac surgery, up to 1000 minutes.
  Cardiopulmonary bypass duration (minutes)
Red blood cells transfusion | Assessed at the end of hospitalization, through study completion, assessed up to 24 months.
  Red blood cells transfusion (units)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Nguyen, MD, MSc, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Bignami E, Guarnieri M, Saglietti F, Belletti A, Trumello C, Giambuzzi I, Monaco F, Alfieri O. Mechanical Ventilation During Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2016 Dec;30(6):1668-1675. doi: 10.1053/j.jvca.2016.03.015. Epub 2016 Mar 9. No abstract available. PMID 27468893
- [Background] Schreiber JU, Lance MD, de Korte M, Artmann T, Aleksic I, Kranke P. The effect of different lung-protective strategies in patients during cardiopulmonary bypass: a meta-analysis and semiquantitative review of randomized trials. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):448-54. doi: 10.1053/j.jvca.2012.01.034. Epub 2012 Mar 28. PMID 22459933
- [Derived] Nguyen LS, Estagnasie P, Merzoug M, Brusset A, Law Koune JD, Aubert S, Waldmann T, Naudin C, Grinda JM, Gibert H, Squara P. Low Tidal Volume Mechanical Ventilation Against No Ventilation During Cardiopulmonary Bypass in Heart Surgery (MECANO): A Randomized Controlled Trial. Chest. 2021 May;159(5):1843-1853. doi: 10.1016/j.chest.2020.10.082. Epub 2020 Nov 17. PMID 33217416
- [Derived] Nguyen LS, Merzoug M, Estagnasie P, Brusset A, Law Koune JD, Aubert S, Waldmann T, Grinda JM, Gibert H, Squara P. Low tidal volume mechanical ventilation against no ventilation during cardiopulmonary bypass heart surgery (MECANO): study protocol for a randomized controlled trial. Trials. 2017 Dec 2;18(1):582. doi: 10.1186/s13063-017-2321-9. PMID 29197407
- See also: Center of Disease Control pneumonia criteria, 2016 update — https://www.cdc.gov/nhsn/PDFs/pscManual/6pscVAPcurrent.pdf